CLINICAL TRIAL: NCT03805256
Title: Preoperative and Postoperative ctDNA Comparison in Early Stage Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: 12345
Record Dates: First submitted 2019-01-12; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Preoperative and Postoperative ctDNA Comparison in Early Stage Lung Cnacer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mutation-positive peripheral blood ctDNA became mutation-negative after surgical removal of the cancer tissue. All subjects in the control group were negative for ctDNA mutations。

ELIGIBILITY:
Inclusion Criteria:Patients with pulmonary nodules who underwent curative-intent resection were able to enter the study -

Exclusion Criteria:Patients who received any invasive examination or treatment prior to resection or had a history of malignancy; patients who do not attend follow up after surgery; blood samples that were contaminated; and biopsies that exhibited advanced lung cancer in pathology。

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population comprises all adult patients aged 18 years and older who present with pulmonary nodules.The study sample will include 60 subjects.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
The potential value of ctDNA in the diagnosis of NSCLC | Half a year
  The sensitivity,specificity,positive predictive valueand the negative predictive value of mutations in plasma ctDNA for detecting early-stage lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Gong, Doctor, Study Director — Second Affiliated Hospital of Soochow University
Locations (1):
- Jianping Gong, Suzhou, Jiangsu, China